CLINICAL TRIAL: NCT02215213
Title: Assessment of Dose Effectiveness of Vitamin D Supplementation During Pregnancy
Brief Title: Assessment of Dose Effectiveness of Vitamin D Supplementation During Pregnancy- a Dose Comparison Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Sidrah Nausheen, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PF8/0911
Record Dates: First submitted 2014-08-06; First posted 2014-08-13 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Pregnancy
Keywords: Vitamin D; pregnancy; Pakistan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Active Comparator): Arm 1 is receiving vitamin D supplementation in 2000 IU/day ,
  Interventions: Drug: Vitamin D supplement
- Arm 2 intervention group (Active Comparator): Arm 2 is receiving vitamin D supplementation in 4000/IU per day
  Interventions: Drug: Vitamin D supplement
- Arm 3 control group (Active Comparator): Arm 3 is receiving vitamin D supplementation in 400 IU/day
  Interventions: Drug: Vitamin D supplement

INTERVENTIONS:
Drug: Vitamin D supplement — comparison of different dosages of vitamin D
  Other Names: Brand name: Vitamin D3; LOT ID AKUH COMPOUNDING 2305012014
Drug: Vitamin D supplement — comparison of different dosages of vitamin D Supplement
  Other Names: Brand name: Vitamin D3

SUMMARY:
The study is randomized blinded trial of Vitamin D supplementation to pregnant women; the study participants will receive Vitamin D in supplement form. Pregnant women will be individually randomized to three groups receiving a dose of 400, 2000 and 4000 IU/ day till the time of delivery.A blood sample will also be collected from the participant at the time of recruitment /before the starting of the supplementation for the assessment of Calcium, Phosphorus, Alkaline Phosphatase and Vitamin D levels. The second blood sample for vitamin D level to assess vitamin D status will be done after completion of the supplementation phase at the time of delivery (till 48 hours of delivery). The samples will be sent to Aga Khan University laboratory

DETAILED DESCRIPTION:
The investigators hypothesize that Pakistani mothers as darkly pigmented, will require substantially higher oral supplementation with vitamin D to replenish the micronutrient stores and aid to resolve associated maternal and neonatal morbidity due to Vitamin D deficiency. The investigators expect that if vitamin D is supplemented to pregnant women, their newborn infants would inevitably replenish the micronutrient stores and aid to resolve the maternal and neonatal morbidity due to Vitamin D deficiency.This is hospital based double blinded trial, study participants divided into three groups which will receive Vitamin D supplementation in 400, 2000 and 4000 International Units. The group which will receive 400 IUs will be treated as control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 15 - 45 years
* Less than 16 weeks pregnant from Last menstrual period.
* Agree to take part in this study, will be enrolled.

Exclusion Criteria:

* Pregnant women with pre existing type 1 or type II diabetes,
* Pregnant women with pre existing hypertension
* Women with multiple fetuses, babies (twins, triplets)
* Women with fetal anomaly in scan
* Refuse to participate in the study

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
pregnancy out come | At delivery of neonate
  Hypovitaminosis, Pre eclampsia, Preterm labour, preterm birth, low birth weight, Still birth rates.

SECONDARY OUTCOMES:
Prevalence of vitamin D deficiency in pregnant women | at recruitment into study (first trimester)
  Maternal vitamin D deficiency in the target group.

CONTACTS AND LOCATIONS:
Overall Officials: Sidrah Nausheen, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Farrant HJ, Krishnaveni GV, Hill JC, Boucher BJ, Fisher DJ, Noonan K, Osmond C, Veena SR, Fall CH. Vitamin D insufficiency is common in Indian mothers but is not associated with gestational diabetes or variation in newborn size. Eur J Clin Nutr. 2009 May;63(5):646-52. doi: 10.1038/ejcn.2008.14. Epub 2008 Feb 20. PMID 18285809
- [Result] Bodnar LM, Catov JM, Roberts JM, Simhan HN. Prepregnancy obesity predicts poor vitamin D status in mothers and their neonates. J Nutr. 2007 Nov;137(11):2437-42. doi: 10.1093/jn/137.11.2437. PMID 17951482
- [Result] Javaid MK, Crozier SR, Harvey NC, Gale CR, Dennison EM, Boucher BJ, Arden NK, Godfrey KM, Cooper C; Princess Anne Hospital Study Group. Maternal vitamin D status during pregnancy and childhood bone mass at age 9 years: a longitudinal study. Lancet. 2006 Jan 7;367(9504):36-43. doi: 10.1016/S0140-6736(06)67922-1. PMID 16399151
- [Result] Gale CR, Robinson SM, Harvey NC, Javaid MK, Jiang B, Martyn CN, Godfrey KM, Cooper C; Princess Anne Hospital Study Group. Maternal vitamin D status during pregnancy and child outcomes. Eur J Clin Nutr. 2008 Jan;62(1):68-77. doi: 10.1038/sj.ejcn.1602680. Epub 2007 Feb 21. PMID 17311057
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Nausheen S, Habib A, Bhura M, Rizvi A, Shaheen F, Begum K, Iqbal J, Ariff S, Shaikh L, Raza SS, Soofi SB. Impact evaluation of the efficacy of different doses of vitamin D supplementation during pregnancy on pregnancy and birth outcomes: a randomised, controlled, dose comparison trial in Pakistan. BMJ Nutr Prev Health. 2021 Sep 27;4(2):425-434. doi: 10.1136/bmjnph-2021-000304. eCollection 2021. PMID 35028513